CLINICAL TRIAL: NCT02666911
Title: Assessing the Comparability of 2D and 4D Ultrasound Measurements of Human Carpal Tunnel Synovium, Median Nerve and Tendon Displacement
Brief Title: Assessing the Comparability of 2D and 4D Ultrasound Measurements
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Equipment to run the study was not available
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Peter C. Amadio, M.D., Consultant - Hand Surgery, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-008487
Record Dates: First submitted 2016-01-15; First posted 2016-01-28 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Carpal Tunnel
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 4D Ultrasound (Experimental): 4D ultrasound imaging of the carpal tunnel. 20 healthy volunteers between the ages of 18 and 80, who have no history of carpal tunnel syndrome or wrist injury. The same patients will be imaged with both 2D and 4D transducers.
  Interventions: Procedure: 4D Ultrasound
- 2D ultrasound (Active Comparator): 2D ultrasound imaging of the carpal tunnel. 20 healthy volunteers between the ages of 18 and 80, who have no history of carpal tunnel syndrome or wrist injury.The same patients will be imaged with both 2D and 4D transducers.
  Interventions: Procedure: 2D ultrasound

INTERVENTIONS:
Procedure: 4D Ultrasound — Each subject will be imaged lying supine on imaging table with affected arm outstretched on Plexiglass board. An ultrasound scanner equipped with 15L8 linear array transducer will be set to depth of 20-25 mm with a 15MHz image acquisition frequency (for longitudinal and transverse imaging) and the same ultrasound machine equipped with 4D transducer will be used. Ultrasound evaluation will be performed by a sonographer trained in the pertinent image acquisition procedures. The image acquisition frame rate will be maintained at 70Hz, and the image compression will be set to low.
  Arms: 4D Ultrasound
Procedure: 2D ultrasound — Each subject will be imaged lying supine on imaging table with affected arm outstretched on Plexiglass board. An ultrasound scanner equipped with 15L8 linear array transducer will be set to depth of 20-25 mm with a 15MHz image acquisition frequency (for longitudinal and transverse imaging) and the same ultrasound machine equipped with 4D transducer will be used. Ultrasound evaluation will be performed by a sonographer trained in the pertinent image acquisition procedures. The image acquisition frame rate will be maintained at 70Hz, and the image compression will be set to low.
  Arms: 2D ultrasound

SUMMARY:
Investigators will recruit 20 healthy volunteers between the ages of 18 and 80, who have no history of carpal tunnel syndrome or wrist injury. Images will be captured twice, first with the 2D transducer and then with the 4D transducer and compared to images captured with the new 4D transducer, using the same movement data analysis protocols. Investigators will also assess the inter and intrarater reliability of the 4D transducer images, by using two different sonographers, both trained in the technique, measuring the same blinded images on separate occasions, at least two weeks apart. The overall goal of this project is to assess the reliability, or reproducibility, of measurements in normal subjects using a novel 4D ultrasonographic method to characterize the subsynovial connective tissue (SSCT) and detect motion between SSCT, median nerve and tendon motion for the evaluation and diagnosis of patients with disorders affecting the carpal tunnel, especially carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
CTS can be diagnosed in many ways, but there are currently no non-invasive methods to assess the physiology within the carpal tunnel, which may help select treatment and predict treatment outcomes. The investigators have shown in preliminary work that differences in the motion of various structures within the carpal tunnel, including the median nerve, flexor tendons, and SSCT, vary in normal subjects and those with CTS. A clinical trial is already under way to assess conventional ultrasound imaging to predict outcomes of CTS treatments. In this study investigators wish to compare the current ultrasound methods, which involve moving two dimensional images, with a new technology which captures moving images in three dimensions (i.e., four dimensions, or 4D). If successful, a single 4D measurement could replace longitudinal and transverse 2D images, saving time and allowing better understanding of the relationship between displacements in both planes.

ELIGIBILITY:
Inclusion Criteria:

• Healthy Volunteers

Exclusion Criteria:

* Cervical radiculopathy
* Rheumatoid arthritis
* Osteoarthritis
* Flexor tendinitis
* Gout
* Hemodialysis
* Sarcoidosis
* Peripheral nerve disease
* Amyloidosis
* Traumatic injury - same arm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
shear index between SSCT and flexor digitorum superficialis 3 tendon (FDS3) | 1 year
  the relative motion of the SSCT and FDS3 on longitudinal video clips, expressed as a ratio of SSCT/FDS3

SECONDARY OUTCOMES:
motion of the median nerve | 1 year
  on cross sectional images, in mm from starting point, while the wrist is flexed
shape of median nerve | 1 year
  on cross sectional images, both cross sectional area in mm squared, and shape in terms of circularity (X axis divided by Y axis)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Amadio, M.D., Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No